CLINICAL TRIAL: NCT05219292
Title: Impact of a Multidisciplinary Protocol of Respiratory Kinesitherapy and Active Music Therapy on Anxiety, Depression and Pain in Lung Transplant Patients: PPKRMA
Brief Title: Impact of a Multidisciplinary Protocol of Respiratory Kinesitherapy and Active Music Therapy on Anxiety, Depression and Pain in Lung Transplant Patients
Acronym: PPKRMA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1061; 2022-A00056-37 (Other: ANSM)
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Lung Transplant; Pain
Keywords: Lung transplantation; Respiratory kinesitherapy; Active music therapy; Anxiety; Depression; Pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients followed for a recent lung transplant.: Patients will be recruited during the pre-transplant assessment by the physiotherapist, the pneumologist and/or the transplant nurse coordinator. The patient has the hospital stay of the pre-transplantation to give his answer. The protocol starts on arrival in the rehabilitation department.
  Interventions: Other: Active music therapy; Other: Questionnaires

INTERVENTIONS:
Other: Active music therapy — Active music therapy is not a musical learning process. The restrictive character of classical respiratory rehabilitation will be alleviated by the playful aspect and the pleasure generated by the sessions, which will facilitate the commitment of the patients in their post-transplant respiratory rehabilitation.
  The recorder was chosen among other wind instruments for several reasons:
  * Its use is simple,
  * It acts as an oscillating exhalation resistance device that generates a positive expiratory pressure (auto-PEP) produced by this wind instrument allows to obtain conditions similar to the treatment performed by a flutter (classical respiratory rehabilitation), a pressure on the expiratory flow with the obtaining of an oscillating effect during the trills, an increase of the respiratory capacities,
  * The characteristics of the sound it produces (duration, intensity, timbre and frequency) will generate auditory feedback allowing patients to become aware of their breathing patterns.
Other: Questionnaires — We chose the HAD (Hospital Anxiety and Depression Scale) to assess anxiety and depression. This test is a reference test, often used in studies of transplant patients. The results obtained in previous studies allowed us to create our hypotheses.
  To measure pain we chose the visual analogue scale (VAS). This reference test is often used in pain studies. It has the advantage of being simple to perform and easy to understand.
  Quality of life will be assessed using the SF-12 (Short Form 12 Health Survey Questionary). We consider it to be simple and easy for patients to understand.

SUMMARY:
Transplantation remains the last resort to prolong life when the patient reaches the stage of terminal respiratory failure. Lung transplantation improves survival and quality of life compared to medical treatment, at acceptable costs. However, the burden of the lived reality and the direct consequences of the operation have considerable impact. The transplant patient faces extraordinary physical and psychological challenges.

While quality of life and long-term prognosis are significantly improved, psychopathological disorders are common, mainly anxiety disorders. A high prevalence of psychopathological disorders is reported in most retrospective and prospective studies. These are essentially adjustment disorders, with depressive mood and/or anxiety, reactive to the severity of the pre- and postoperative somatic reality.

The partial or total replacement of the respiratory "bellows" leads to more anxiety disorders than in other transplants. Quality of life is a multidimensional concept that encompasses medical, social, cultural, psychological and economic factors. It is based on four dimensions: physical state, somatic sensations, psychological state, social status. Regarding the quality of psychic evolution after transplantation, among the criteria that are usually analysed we find adaptation to body changes and anxiety management.

Meta-analyses of clinical trials have shown that music therapy, which is based on the use of the properties of music and sound for therapeutic purposes, has an impact on the human being, reducing anxiety, depression and pain. Two clinical trials have shown that pulmonary rehabilitation with active music therapy improves lung function and reduces dyspnoea. The concept of active music therapy, which emphasises sound production and improvisation, is a controlled technique of musical practice for therapeutic purposes. Playing a wind instrument, using vocal techniques and respiratory rhythm modulation techniques, would provide additional benefits for respiratory function.

The use of recorders as an oscillating exhalation resistance device will provide conditions similar to the treatment provided by a flutter, a device that creates exhalation resistance and improves secretion clearance.

Investigators hypothesize that the combination of Respiratory Kinesitherapy and active breath music therapy (PPKRMA) will address anxiety, depression, and pain in lung.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged at least 18 years and less than 70 years.
* Patient who has had a lung transplant for less than 5 weeks and who has been transferred to the participating department that provides post-transplant follow-up.
* Patient who has completed the pre-transplant assessment according to the practices of the receiving department.
* Clinically stable as judged by the investigator (pulmonologist).
* Patient who has been informed of the study and has given his agreement to participate.

Exclusion Criteria:

* Impaired perception of music as judged by the investigator: musicogenic epilepsy (i.e. seizures provoked by music), hyperacusis (i.e. an abnormally low threshold of tolerance to noise), dysmusia (music is perceived as an annoying noise), amusia (rhythm, melody, chords of music are not perceived) .
* Physical inability to perform the PPKRMA.
* Neurocognitive disorders that do not allow the PPKRMA, the questionnaires required by the protocol or the functional explorations to be carried out.
* Dependence on oxygen therapy with a flow rate of more than 5l of O2.
* Persons deprived of liberty by judicial or administrative decision
* Persons subject to psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Persons of full age subject to a legal protection measure (guardianship, curatorship).
* Subjects participating in other interventional research with an exclusion period still in progress at pre-inclusion or which may interfere with the results of this research protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during the pre-transplant assessment by the physiotherapist, the pneumologist and/or the transplant nurse coordinator. The patient has the hospital stay of the pre-transplantation to give his answer. The protocol starts on arrival in the rehabilitation department.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Evolution of anxiety | 28 days
  Evolution of anxiety with the HAD (Hospital Anxiety and Depression) scale scores between the beginning and the end of the treatment in the rehabilitation service.
Evolution of depression | 28 days
  Evolution of depression with the HAD (Hospital Anxiety and Depression) scale) scores between the beginning and the end of the treatment in the rehabilitation service.
Evolution of pain | 28 days
  Evolution of pain with the visual analogue scale (VAS) scores between the beginning and the end of the treatment in the rehabilitation service

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumologie C Bât A4 Hôpital cardiologique Louis Pradel, Groupement Hospitalier Est Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No